CLINICAL TRIAL: NCT06884579
Title: Educational Programs Based on Healthy Habits to Improve Quality of Life and Psychosocial Profile in Women With Neurodegenerative Diseases: The ADVICE Protocol Study
Brief Title: Educational Programs Based on Healthy Habits to Improve Quality of Life and Psychosocial Profile in Women With Neurodegenerative Diseases: the ADVICE Protocol Study (Phase 2)
Acronym: ADVICE Phase 2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Hospital Universitario Virgen de la Arrixaca (Other)
Responsible Party: Principal Investigator, Jacobo Á. Rubio-Arias, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-3-15-HCUVA; PID2021-123447OA-I00 (Other: MCIN/AEI /10.13039/501100011033 and by FEDER, UE.)
Record Dates: First submitted 2025-02-20; First posted 2025-03-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS) - Relapsing-remitting
Keywords: Relapsing-Remitting MS; Fatigue; Cognitive Behavioral Therapy; Physical exercise; Dietary habits; Women's Health
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Fatigue; Motor Activity; Feeding Behavior | interventions — Resistance Training; Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supervised Strength Training Program (PE1) (Experimental): Participants will complete 36 strength sessions (3 times a week) at a moderate intensity, 6 educational nutritional intervention sessions, and 8 sessions on energy and fatigue management.
  Interventions: Other: Strength training, nutrition, and behavioral training
- Self-Guided and Unsupervised Program with General Recommendations (PE1) (Active Comparator): Participants will be involved in an unsupervised, self-directed program focusing on physical exercise (three times per week), nutrition and cognitive-behavioral habits.
  Interventions: Other: Self-Guided and Unsupervised Program with General Recommendations

INTERVENTIONS:
Other: Strength training, nutrition, and behavioral training — This arm of the study consists of a supervised strength training program, conducted over 12 weeks with three weekly sessions. The sessions follow a wave-like periodization, with intensities ranging from 70% to 85% of 1-RM. Exercises focus on enhancing neuromuscular strength in the lower limbs, such as leg presses and hip extensions, under the supervision of a multidisciplinary team.
  Participants will also receive nutritional guidance based on the Mediterranean diet, as well as cognitive-behavioral therapy strategies aimed at optimizing fatigue management and boosting energy levels.
  Arms: Supervised Strength Training Program (PE1)
Other: Self-Guided and Unsupervised Program with General Recommendations — This arm of the study consists of a self-guided and unsupervised program based on physical exercise (3 times per week), nutrition, and cognitive-behavioral habits. Participants will access online modules that provide guidelines for performing resistance exercises with bands, dietary recommendations following the principles of the Mediterranean diet, and cognitive-behavioral techniques for fatigue management.
  Arms: Self-Guided and Unsupervised Program with General Recommendations (PE1)

SUMMARY:
This phase of the project aims to compare in-person, supervised educational programs (EP) with online self-guided EPs in individuals with relapsing-remitting multiple sclerosis. A total of 75 participants will be randomly assigned to one of three groups: a supervised and individualized educational program focused on HIIT training, a supervised and individualized educational program focused on strength training, and a non-supervised, self-guided educational program based on resistance band training. Additionally, sessions on the Mediterranean diet (both supervised and non-supervised) and cognitive-behavioral interventions will be included. A control evaluation will be conducted three months after the intervention to assess the effects of the educational programs, followed by another evaluation three months later to analyze residual effects. Women who participated in Phase 1 of the study will be invited to take part in this second phase.

ELIGIBILITY:
Inclusion criteria include:

* Women and men of reproductive age (18-45 years) with MS will be included, with the upper age limit adjusted to reflect the reproductive phase;
* no iron-deficiency anemia;
* stable disease phase;
* independent walking ability for over 10 meters.

Women will be recruited first and later matched with men based on age, EDSS, and lifestyle habits (physical activity, smoking, and alcohol consumption).

Exclusion criteria will include participants with MS who:

* score <1 or >6 on the EDSS;
* report a relapse within 12 months before the study begins;
* have taken corticosteroid treatment within the last 2 months;
* have participated in a structured training program in the previous 6 months.

Once all women with MS are recruited, male participants will be recruited following a 1:1 matching methodology based on age, geographic region, and lifestyle habits.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Physical Activity | Baseline (pre-intervention)
  Satisfaction with Physical Activity will be measured using an eight-item, 5-point Likert scale
Satisfaction with Physical Activity | Immediately after the intervention
  Satisfaction with Physical Activity will be measured using an eight-item, 5-point Likert scale
Visual Analogue Scale for Fatigue (VAS-F) | Immediately before each of the 36 exercise sessions (pre-session assessment).
  The Visual Analogue Scale for Fatigue (VAS-F) assesses subjective levels of fatigue and energy
Visual Analogue Scale for Fatigue (VAS-F) | Immediately after each of the 36 exercise sessions (post-session assessment).
  The Visual Analogue Scale for Fatigue (VAS-F) assesses subjective levels of fatigue and energy
Modified Fatigue Impact Scale (MFIS) | Baseline (pre-intervention).
  Fatigue perception will be measured using the MFIS. This scale is a 21-item multidimensional questionnaire that evaluates the physical, cognitive, and psychosocial effects of fatigue on a five-point ordinal scale (with a maximum total score of 84).
Modified Fatigue Impact Scale (MFIS) | 48 hours after the last exercise session (post-intervention assessment).
  Fatigue perception will be measured using the MFIS. This scale is a 21-item multidimensional questionnaire that evaluates the physical, cognitive, and psychosocial effects of fatigue on a five-point ordinal scale (with a maximum total score of 84)

SECONDARY OUTCOMES:
Inflammatory Profile | Baseline (pre-intervention).
  The inflammatory profile evaluates key cytokines, including IFN-γ, IL-6, TNF-α, IL-10, and TGF-β1, to assess systemic inflammation and immune response dynamics
Inflammatory Profile | 48 hours after the last exercise session (post-intervention assessment).
  The inflammatory profile evaluates key cytokines, including IFN-γ, IL-6, TNF-α, IL-10, and TGF-β1, to assess systemic inflammation and immune response dynamics
The hormonal profile | Pre-intervention in each phase of the menstrual cycle (early follicular phase, late follicular phase and mid-luteal phase).
  The hormonal profile includes the assessment of TSH, progesterone (PG), luteinizing hormone (LH), follicle-stimulating hormone (FSH), estradiol, and testosterone to evaluate endocrine function, menstrual cycle phases, and hormonal balance.
Cognitive Function | Baseline (pre-intervention).
  Brain-Derived Neurotrophic Factor (BDNF) is a protein involved in neuroplasticity, cognitive function, and neuronal survival, serving as a blood biomarker for brain health and adaptability.
Cognitive Function | 48 hours after the last exercise session (post-intervention assessment).
  Brain-Derived Neurotrophic Factor (BDNF) is a protein involved in neuroplasticity, cognitive function, and neuronal survival, serving as a blood biomarker for brain health and adaptability
Neurofilament Light Chain (NFL) | Baseline (pre-intervention).
  Neurofilament light chain (NFL) is one of the most relevant biomarkers in multiple sclerosis (MS). The Simoa detection technique (ultrasensitive single-molecule array) allows its analysis in serum, providing both the total value and the Z-Score, enabling precise assessment of axonal damage and disease progression.
Neurofilament Light Chain (NFL) | 48 hours after the last exercise session (post-intervention assessment).
  Neurofilament light chain (NFL) is one of the most relevant biomarkers in multiple sclerosis (MS). The Simoa detection technique (ultrasensitive single-molecule array) allows its analysis in serum, providing both the total value and the Z-Score, enabling precise assessment of axonal damage and disease progression.
Physical Self-Perception | Baseline (pre-intervention).
  Physical self-perception will be evaluated using six subscales-sports competence, physical condition, body attractiveness, physical strength, general physical self-perception, and overall self-perception-on a 5-point Likert scale
Physical Self-Perception | 48 hours after the last exercise session (post-intervention assessment).
  Physical self-perception will be evaluated using six subscales-sports competence, physical condition, body attractiveness, physical strength, general physical self-perception, and overall self-perception-on a 5-point Likert scale
Walking Endurance | Baseline (pre-intervention).
  Participants will undergo the 2-minute walk test, during which they will walk at their preferred, self-selected speed to assess walking endurance. The test course will be rectangular, with corners marked by cones. Participants will be allowed to rest during the test, if necessary, but the clock will not stop during these rest periods. The total distance covered will be recorded
Walking Endurance | 48 hours after the last exercise session (post-intervention assessment).
  Participants will undergo the 2-minute walk test, during which they will walk at their preferred, self-selected speed to assess walking endurance. The test course will be rectangular, with corners marked by cones. Participants will be allowed to rest during the test, if necessary, but the clock will not stop during these rest periods. The total distance covered will be recorded
Pain Catastrophizing | Baseline (pre-intervention).
  The Pain Catastrophizing Scale will measure catastrophic thoughts related to pain, focusing on rumination and helplessness, with responses on a similar scale
Pain Catastrophizing | 48 hours after the last exercise session (post-intervention assessment).
  The Pain Catastrophizing Scale will measure catastrophic thoughts related to pain, focusing on rumination and helplessness, with responses on a similar scale
Quality of Life questionnaire | Baseline (pre-intervention).
  The Multiple Sclerosis Quality of Life-54 will gauge quality of life across 14 subscales, yielding physical and mental health composite scores
Quality of Life questionnaire | 48 hours after the last exercise session (post-intervention assessment).
  The Multiple Sclerosis Quality of Life-54 will gauge quality of life across 14 subscales, yielding physical and mental health composite scores
State-Trait Anxiety | Baseline (pre-intervention).
  Description: The State-Trait Anxiety Inventory will measure both situational and general anxiety on a 4-point scale
State-Trait Anxiety | 48 hours after the last exercise session (post-intervention assessment).
  The State-Trait Anxiety Inventory will measure both situational and general anxiety on a 4-point scaleTime Frame: Before the first training session
Rate of force development | Baseline (pre-intervention).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). They will perform three maximum contractions, each lasting 2 seconds, with 3 minutes of rest in between. The RFD will be analyzed. Testing will begin with the right leg, and the repetition with the highest recorded value for each leg will be used in the analysis
Rate of force development | 48 hours after the last exercise session (post-intervention assessment).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway). They will perform three maximum contractions, each lasting 2 seconds, with 3 minutes of rest in between. The RFD will be analyzed. Testing will begin with the right leg, and the repetition with the highest recorded value for each leg will be used in the analysis
Maximum Voluntary Isometric Contraction | Baseline (pre-intervention).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway).Participants will perform three 5-second MVIC, with 3 minutes of rest in between. Testing will always begin with the right leg, and the contraction with the highest recorded MVIC value will be used in the analysis Time Frame: Before the first training session
Maximum Voluntary Isometric Contraction | 48 hours after the last exercise session (post-intervention assessment).
  Participants will sit in a chair with both legs flexed at a 90-degree angle, and the tested ankle securely attached to a customized device with a load cell (MuscleLab Force Sensor, Ergotest AS, Langesund, Norway).Participants will perform three 5-second MVIC, with 3 minutes of rest in between. Testing will always begin with the right leg, and the contraction with the highest recorded MVIC value will be used in the analysis Time Frame: Before the first training session
Maximal neural drive | Baseline (pre-intervention).
  To measure neural drive, the electromyographic activity (sEMG) of the right leg's vastus lateralis will be recorded during the MVIC (Delsys Trigno, Delsys Inc., Boston, MA) with skin prepared and electrode positioning following SENIAM guidelines. EMG peak will be analyzed. The EMG peak during MVIC will represent the maximum neural drive
Maximal neural drive | 48 hours after the last exercise session (post-intervention assessment).
  To measure neural drive, the electromyographic activity (sEMG) of the right leg's vastus lateralis will be recorded during the MVIC (Delsys Trigno, Delsys Inc., Boston, MA) with skin prepared and electrode positioning following SENIAM guidelines. EMG peak will be analyzed. The EMG peak during MVIC will represent the maximum neural drive
Central activation ratio | Baseline (pre-intervention).
  Two bipolar electrodes (10×15 cm) will be placed on the right quadriceps, with electrical stimulation controlled by Signal 6.0 software (CED, Cambridge, England) at 100 Hz frequency, 50 pulses, 0.009 s pulse duration, and 0.01 s interval, set to 40-50% of MVIC. Central activation ratio (CAR) will be assessed through a sequence of one supramaximal twitch, a 100 Hz tetanic train, an MVIC with superimposed tetanic train, followed by a potentiated tetanic train and a potentiated supramaximal twitch. This sequence will be repeated twice with 2-minute rests, and twitch-to-tetanus ratio, MVIC peak, and maximum force values will be calculated for CAR. The CAR will be calculated using the following formula: "CAR= " "Force during MVIC" /"Force during MVIC + supramaximal stimulation"
Central activation ratio | 48 hours after the last exercise session (post-intervention assessment).
  Two bipolar electrodes (10×15 cm) will be placed on the right quadriceps, with electrical stimulation controlled by Signal 6.0 software (CED, Cambridge, England) at 100 Hz frequency, 50 pulses, 0.009 s pulse duration, and 0.01 s interval, set to 40-50% of MVIC. Central activation ratio (CAR) will be assessed through a sequence of one supramaximal twitch, a 100 Hz tetanic train, an MVIC with superimposed tetanic train, followed by a potentiated tetanic train and a potentiated supramaximal twitch. This sequence will be repeated twice with 2-minute rests, and twitch-to-tetanus ratio, MVIC peak, and maximum force values will be calculated for CAR. The CAR will be calculated using the following formula: "CAR= " "Force during MVIC" /"Force during MVIC + supramaximal stimulation"
Upper Limb Maximum Strength | Baseline (pre-intervention).
  Isometric grip strength will be measured with an electronic dynamometer (K-Force Grip, Kinvent, Montpellier, France) as participants stand with elbows extended. Each hand will perform 3 trials, with 30 seconds rest between attempts
Upper Limb Maximum Strength | 48 hours after the last exercise session (post-intervention assessment).
  Isometric grip strength will be measured with an electronic dynamometer (K-Force Grip, Kinvent, Montpellier, France) as participants stand with elbows extended. Each hand will perform 3 trials, with 30 seconds rest between attempts
Spasticity | Before the first session of the intervention program
  The Pendulum Test is used to assess the level of spasticity by evaluating the resistance to passive movement in the affected limb. The test involves moving the limb in a pendulum-like motion and observing the fluidity of the movement, with increased resistance indicating higher spasticity levels
Spasticity | 48 hours after the last exercise session (post-intervention assessment).
  The Pendulum Test is used to assess the level of spasticity by evaluating the resistance to passive movement in the affected limb. The test involves moving the limb in a pendulum-like motion and observing the fluidity of the movement, with increased resistance indicating higher spasticity levels
Intrinsic muscle characteristics | Baseline (pre-intervention).
  Muscle characteristics (frequency, stiffness, degradation) assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia)
Intrinsic muscle characteristics | 48 hours after the last exercise session (post-intervention assessment).
  Muscle characteristics (frequency, stiffness, degradation) assessed with MyotonPRO (MyotonPRO, Myoton AS, Estonia)
Gait speed | Baseline (pre-intervention).
  Gait speed will be determined with the 10-meter walk test using two photocells (Ergotest Technology AS, Langesund, Norway) at 5 and 10 meters; participants will complete two maximum-speed trials, with the slower time recorded
Gait speed | 48 hours after the last exercise session (post-intervention assessment).
  Gait speed will be determined with the 10-meter walk test using two photocells (Ergotest Technology AS, Langesund, Norway) at 5 and 10 meters; participants will complete two maximum-speed trials, with the slower time recorded
Static balance with eyes open | Baseline (pre-intervention).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Static balance with eyes open | 48 hours after the last exercise session (post-intervention assessment).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Static balance with eyes closed | Baseline (pre-intervention).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Static balance with eyes closed | 48 hours after the last exercise session (post-intervention assessment).
  Balance is measured with static trials on a force platform (Ergotest Technology AS, Langesund, Norway), where participants stand barefoot with arms at their sides for two 30-second trials each
Sit-to-stand | Baseline (pre-intervention).
  The sit-to-stand test requires participants to rise as quickly as possible from a seated position with 90º knee flexion and arms crossed
Sit-to-stand | 48 hours after the last exercise session (post-intervention assessment).
  The sit-to-stand test requires participants to rise as quickly as possible from a seated position with 90º knee flexion and arms crossed
Timed Up-and-Go test | Baseline (pre-intervention).
  In the Timed Up-and-Go test, participants move from sitting to standing, walk 3 meters, turn, return, and sit
Timed Up-and-Go test | 48 hours after the last exercise session (post-intervention assessment).
  In the Timed Up-and-Go test, participants move from sitting to standing, walk 3 meters, turn, return, and sit
Delayed onset muscle soreness | Baseline (pre-intervention).
  To measure delayed onset muscle soreness (DOMS), a 10-point visual analogue scale shall be used, where 1 = no pain and 10 = intolerable pain
Subjective Perception of Effort | Baseline (pre-intervention).
  Participants will be instructed and familiarized with the use of the RPE scale during the familiarization phase. RPE will be assessed before, during (after each exercise within the session), and after the training session using the Borg 6-20 RPE scale
Fatigue Visual Analog Scale (VAS-F) | Baseline (pre-intervention).
  The VAS-F will be used to measure fatigue. This scale, is subdivided into two subscales: fatigue and energy. The VAS-F features a 100 mm long horizontal line, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line corresponding to their perception of the severity of fatigue between these two endpoints.
Anthropometric | Baseline (pre-intervention).
  Anthropometric measurements will be taken to assess body morphology, fat distribution, and potential alterations due to multiple sclerosis (MS), such as muscle atrophy or changes in body fat percentage. These measurements provide valuable information regarding comorbidities, including abdominal obesity and cardiovascular risk, which are particularly relevant in MS due to factors like reduced mobility or medication use
Anthropometric | 48 hours after the last exercise session (post-intervention assessment).
  Anthropometric measurements will be taken to assess body morphology, fat distribution, and potential alterations due to multiple sclerosis (MS), such as muscle atrophy or changes in body fat percentage. These measurements provide valuable information regarding comorbidities, including abdominal obesity and cardiovascular risk, which are particularly relevant in MS due to factors like reduced mobility or medication use
Bioimpedance | Baseline (pre-intervention).
  Bioimpedance will be used to assess body composition, including body fat percentage, lean mass, and total body water. These measurements are important for understanding changes in body composition due to multiple sclerosis (MS), as the disease can impact muscle mass, fluid balance, and fat distribution. Bioimpedance provides valuable insight into the health status and nutritional needs of individuals with MS
Bioimpedance | 48 hours after the last exercise session (post-intervention assessment).
  Bioimpedance will be used to assess body composition, including body fat percentage, lean mass, and total body water. These measurements are important for understanding changes in body composition due to multiple sclerosis (MS), as the disease can impact muscle mass, fluid balance, and fat distribution. Bioimpedance provides valuable insight into the health status and nutritional needs of individuals with MS
Physical Activity Levels | Baseline (pre-intervention).
  To assess physical activity in patients with multiple sclerosis (MS), both the International Physical Activity Questionnaire (IPAQ) and triaxial accelerometers can be adapted to account for the mobility limitations often experienced by these individuals. The IPAQ can be tailored by including questions that specifically address low-impact or moderate-intensity activities, considering factors such as fatigue and muscle weakness. Triaxial accelerometers, which measure movement in three planes (vertical, lateral, and anterior-posterior), provide a more detailed and precise measurement of physical activity, capturing even small movements or low-intensity activities such as walking short distances. Together, these tools allow for a comprehensive assessment of physical activity levels in MS patients, while considering their unique needs and capabilities. Additionally, the MET (Metabolic Equivalent of Task) methodology should be adjusted to reflect the lower intensity of activities commonly p
Physical Activity Levels | 48 hours after the last exercise session (post-intervention assessment).
  To assess physical activity in patients with multiple sclerosis (MS), both the International Physical Activity Questionnaire (IPAQ) and triaxial accelerometers can be adapted to account for the mobility limitations often experienced by these individuals. The IPAQ can be tailored by including questions that specifically address low-impact or moderate-intensity activities, considering factors such as fatigue and muscle weakness. Triaxial accelerometers, which measure movement in three planes (vertical, lateral, and anterior-posterior), provide a more detailed and precise measurement of physical activity, capturing even small movements or low-intensity activities such as walking short distances. Together, these tools allow for a comprehensive assessment of physical activity levels in MS patients, while considering their unique needs and capabilities. Additionally, the MET (Metabolic Equivalent of Task) methodology should be adjusted to reflect the lower intensity of activities commonly p
Dietary and Nutritional Follow-up | Baseline (pre-intervention).
  Mediterranean Diet adherence questionnaires and food diaries could be effective tools for evaluating nutrition, particularly if MS patients have poor consumption of essential nutrients for their overall health
Dietary and Nutritional Follow-up | 48 hours after the last exercise session (post-intervention assessment).
  Mediterranean Diet adherence questionnaires and food diaries could be effective tools for evaluating nutrition, particularly if MS patients have poor consumption of essential nutrients for their overall health
The Kurtzke Disability Scale | Baseline (pre-intervention).
  The Kurtzke Disability Scale (EDSS) is divided into 8 functional systems (FS); four primary: pyramidal function, cerebellar function, sensory function, and brainstem function; and four secondary: sphincters, vision, mental, and others. For each FS, a severity score is provided, ranging from 0 to 6 or 7. The overall score of the scale is measured on a 20-item scale (from 0 to 10 points, increasing in half-point increments). Up to 3.5, the score obtained in each FS and the number of affected FS automatically determine the EDSS score. From 4 to 7, the definition of each level is also given by the ability to walk (ability to walk without stopping, need for assistance)
The Kurtzke Disability Scale | 48 hours after the last exercise session (post-intervention assessment).
  The Kurtzke Disability Scale (EDSS) is divided into 8 functional systems (FS); four primary: pyramidal function, cerebellar function, sensory function, and brainstem function; and four secondary: sphincters, vision, mental, and others. For each FS, a severity score is provided, ranging from 0 to 6 or 7. The overall score of the scale is measured on a 20-item scale (from 0 to 10 points, increasing in half-point increments). Up to 3.5, the score obtained in each FS and the number of affected FS automatically determine the EDSS score. From 4 to 7, the definition of each level is also given by the ability to walk (ability to walk without stopping, need for assistance).
Subjective Sleep Quality Questionnaire | Baseline (pre-intervention).
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnaire [73]. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (woke up too early [1] - did not wake up early [3]), e) ease of waking up (very difficult [1] - very easy [5]), f) feeling of rest (did not rest at all [1] - fully rested [3]), and g) sufficient sleep (no, definitely too little [1] - yes, definitely enough [5]).
Subjective Sleep Quality Questionnaire | 48 hours after the last exercise session (post-intervention assessment).
  Subjective sleep quality will be measured using the Karolinska Sleep Diary questionnaire [73]. The questionnaire includes the following items: a) sleep quality (very poor [1] - very good [5]), b) sleep tranquility (very restless [1] - very calm [5]), c) ease of falling asleep (very difficult [1] - very easy [5]), d) awakenings (woke up too early [1] - did not wake up early [3]), e) ease of waking up (very difficult [1] - very easy [5]), f) feeling of rest (did not rest at all [1] - fully rested [3]), and g) sufficient sleep (no, definitely too little [1] - yes, definitely enough [5]).
Sleep Quality Measured by Actigraph | The week prior to the start of the intervention. Baseline (pre-intervention).
  Sleep quality based on actigraphy will be evaluated using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK) [74]. This device uses a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower sensitivity threshold for actigraphy will be set at 80 counts/epoch. Data analysis will begin at the start of the nighttime rest period (bedtime) and conclude at the start of daytime activity (wake-up time).
Sleep Quality Measured by Actigraph | The week following the completion of the intervention (post-intervention assessment).
  Sleep quality based on actigraphy will be evaluated using the Actiwatch wGT3X-BT activity monitoring system (Cambridge Neurotechnology, Cambridge, UK) [74]. This device uses a piezoelectric accelerometer to measure activity. Participants will wear the Actiwatch on their non-dominant wrist. The lower sensitivity threshold for actigraphy will be set at 80 counts/epoch. Data analysis will begin at the start of the nighttime rest period (bedtime) and conclude at the start of daytime activity (wake-up time)
Delayed onset muscle soreness | Immediately after each physical exercise session (post-intervention assessment).
  To measure delayed onset muscle soreness (DOMS), a 10-point visual analogue scale shall be used, where 1 = no pain and 10 = intolerable pain
Subjective Perception of Effort | Immediately after each physical exercise session (post-intervention assessment).
  Participants will be instructed and familiarized with the use of the RPE scale during the familiarization phase. RPE will be assessed before, during (after each exercise within the session), and after the training session using the Borg 6-20 RPE scale
Fatigue Visual Analog Scale (VAS-F) | Immediately after each physical exercise session (post-intervention assessment).
  The VAS-F will be used to measure fatigue. This scale, is subdivided into two subscales: fatigue and energy. The VAS-F features a 100 mm long horizontal line, with the term "none" at one end and "very severe" at the opposite end. Participants are required to mark the point on the line corresponding to their perception of the severity of fatigue between these two endpoints.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Virgen de la Arrixaca, Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided